CLINICAL TRIAL: NCT03140527
Title: A Multi-Center, Randomized, Placebo-Controlled, Phase 1, Two-Part Study Designed to Assess the Safety, Tolerability, Pharmacokinetics, Food Effect, and Drug-Drug Interactions of PTI-801 in Healthy Volunteers, and Safety, Tolerability, and Pharmacokinetics of PTI-801 in Subjects With Cystic Fibrosis
Brief Title: Study Assessing the Safety, Tolerability, Pharmacokinetics, Food Effect, and Drug-Drug Interactions of PTI-801 in Healthy Volunteers, and Safety, Tolerability, and Pharmacokinetics of PTI-801 in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PTI-801-01
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteer; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- SAD HV PTI-801 Active - Complete (Active Comparator): The safety, tolerability, and pharmacokinetic profile of PTI-801 will be evaluated following a single dose of PTI-801. Three cohorts are planned for evaluation where subjects will be randomized to PTI-801 or placebo.The subjects will be followed for 7 days post dose.
  Interventions: Drug: PTI-801
- SAD HV PTI-801 Placebo - Complete (Placebo Comparator): The safety, tolerability, and pharmacokinetic profile of PTI-801 will be evaluated following a single dose of PTI-801. Three cohorts are planned for evaluation where subjects will be randomized to PTI-801 or placebo.The subjects will be followed for 7 days post dose.
  Interventions: Drug: Placebo
- MAD HV PTI-801 Active - Complete (Active Comparator): Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to either PTI-801 or placebo. Each dose will be administered once daily (QD) for a total of 7 days. Follow up visits will occur on Days 10, 12 and 14.
  Interventions: Drug: PTI-801
- MAD HV PTI-801 Placebo - Complete (Placebo Comparator): Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to either PTI-801 or placebo. Each dose will be administered once daily (QD) for a total of 7 days. Follow up visits will occur on Days 10, 12 and 14.
  Interventions: Drug: Placebo
- FE HV PTI-801 Active - Complete (Active Comparator): Following the conclusion of SAD groups and after sufficient review of study data and approval by the SRC, a third set of healthy adult subjects will participate in the Food Effect cohort. Subjects will be randomized to Fed or Fasted on Days 1 and 12. Follow up visits will occur 7 days post Day 12 dose.
  Interventions: Drug: PTI-801
- DDI HV PTI-801 Active - Complete (Active Comparator): Following the conclusion of HV MAD Cohort 2 and after sufficient review of study data and approval by the SRC, a fourth set of healthy adult subjects will participate in the Drug-Drug Interactions cohort. Subjects will receive a 3-drug cocktail consisting of caffeine, bupropion, and midazolam on Day 1. On Day 4, subjects will be randomized to receive either PTI-801 or placebo QD for a total of 12 days. On Day 17, subjects will receive the 3-drug cocktail in combination with PTI-801 or placebo. Subjects will remain in clinic until Day 20. A follow up visit will occur on Day 24.
  Interventions: Drug: PTI-801
- DDI HV PTI-801 Placebo - Complete (Placebo Comparator): Following the conclusion of HV MAD Cohort 2 and after sufficient review of study data and approval by the SRC, a fourth set of healthy adult subjects will participate in the Drug-Drug Interactions cohort. Subjects will receive a 3-drug cocktail consisting of caffeine, bupropion, and midazolam on Day 1. On Day 4, subjects will be randomized to receive either PTI-801 or placebo QD for a total of 12 days. On Day 17, subjects will receive the 3-drug cocktail in combination with PTI-801 or placebo. Subjects will remain in clinic until Day 20. A follow up visit will occur on Day 24.
  Interventions: Drug: Placebo
- MAD Cohort 1-3 CF PTI-801 Active - Complete (Active Comparator): Adult subjects diagnosed with CF currently on stable ivacaftor/lumacaftor background therapy for a minimum of three months will participate in the Part 2 complementary CF MAD cohort. The CF MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to receive either PTI-801 or placebo QD for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: PTI-801
- MAD Cohort 1-3 CF PTI-801 Placebo - Complete (Placebo Comparator): Adult subjects diagnosed with CF currently on stable ivacaftor/lumacaftor background therapy for a minimum of three months will participate in the Part 2 complementary CF MAD cohort. The CF MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to receive either PTI-801 or placebo QD for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: Placebo
- Cohort 4 CF PTI-801 Active co-admin PTI-808 Active - Complete (Active Comparator): Adult subjects diagnosed with CF not currently receiving a CFTR modulator therapy within 30 days prior to Day 1 will participate in the Part 2 CF Cohort 4. Subjects will be randomized to receive either PTI-801 co-administered with PTI-808 or placebos QD.
  Interventions: Drug: PTI-801; Drug: PTI-808
- Cohort 4 CF PTI-801 Placebo co-admin PTI-808 Placebo- Complete (Placebo Comparator): Adult subjects diagnosed with CF not currently receiving a CFTR modulator therapy within 30 days prior to Day 1 will participate in the Part 2 CF Cohort 4. Subjects will be randomized to receive either PTI-801 co-administered with PTI-808 or placebos QD.
  Interventions: Drug: Placebo
- Cohort 5 CF PTI-801 Active co-admin with PTI-808 Active (Active Comparator): Adult subjects diagnosed with CF not currently receiving a CFTR modulator therapy within 30 days prior to Day 1 will participate in the Part 2 CF Cohort 5. Subjects will be randomized to receive either PTI-801 co-administered with PTI-808 or placebos QD.
  Interventions: Drug: PTI-801; Drug: PTI-808
- Cohort 5 CF PTI-801 Placebo co-admin with PTI-808 Placebo (Placebo Comparator): Adult subjects diagnosed with CF not currently receiving a CFTR modulator therapy within 30 days prior to Day 1 will participate in the Part 2 CF Cohort 5. Subjects will be randomized to receive either PTI-801 co-administered with PTI-808 or placebos QD.
  Interventions: Drug: Placebo
- Cohort 6 CF PTI-801 Active (Active Comparator): Adult subjects diagnosed with CF currently on stable tezacaftor/ivacaftor background therapy for a minimum of one month will participate in the Part 2 complementary CF MAD cohort. Subjects will be randomized to receive either PTI-801 or placebo QD.
  Interventions: Drug: PTI-801
- Cohort 6 CF PTI-801 Placebo (Placebo Comparator): Adult subjects diagnosed with CF currently on stable tezacaftor/ivacaftor background therapy for a minimum of one month will participate in the Part 2 complementary CF MAD cohort. Subjects will be randomized to receive either PTI-801 or placebo QD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTI-801 — Active
  Arms: Cohort 4 CF PTI-801 Active co-admin PTI-808 Active - Complete; Cohort 5 CF PTI-801 Active co-admin with PTI-808 Active; Cohort 6 CF PTI-801 Active; DDI HV PTI-801 Active - Complete; FE HV PTI-801 Active - Complete; MAD Cohort 1-3 CF PTI-801 Active - Complete; MAD HV PTI-801 Active - Complete; SAD HV PTI-801 Active - Complete
Drug: Placebo — Placebo
  Arms: Cohort 4 CF PTI-801 Placebo co-admin PTI-808 Placebo- Complete; Cohort 5 CF PTI-801 Placebo co-admin with PTI-808 Placebo; Cohort 6 CF PTI-801 Placebo; DDI HV PTI-801 Placebo - Complete; MAD Cohort 1-3 CF PTI-801 Placebo - Complete; MAD HV PTI-801 Placebo - Complete; SAD HV PTI-801 Placebo - Complete
Drug: PTI-808 — Active
  Arms: Cohort 4 CF PTI-801 Active co-admin PTI-808 Active - Complete; Cohort 5 CF PTI-801 Active co-admin with PTI-808 Active
Drug: Placebo — Placebo
  Arms: Cohort 4 CF PTI-801 Placebo co-admin PTI-808 Placebo- Complete; Cohort 5 CF PTI-801 Placebo co-admin with PTI-808 Placebo

SUMMARY:
This trial will consist of two parts: Part 1 and Part 2. Part 1 will enroll adult healthy volunteers (HV) into four treatment groups. The first group will enroll HV into a single ascending dose (SAD) treatment group consisting of three cohorts. The second group will enroll HV into a multiple ascending dose (MAD) treatment group consisting of three cohorts. The third group will enroll HV into a food effect (FE) treatment group consisting of one cohort. The fourth group will enroll HV into a drug-drug interactions (DDI) treatment group consisting of one cohort. Approximately 76 subjects will be enrolled in Part 1.

Part 2 Cohorts 1 through 3 will enroll adult subjects with cystic fibrosis (CF) currently on stable ivacaftor/lumacaftor background therapy for a minimum of three months. Part 2 Cohorts 4 and Cohort 5 will enroll adult subjects with CF not currently receiving cystic fibrosis conductance regulator (CFTR) modulator therapy within 30 days prior to Day 1. Part 2 Cohort 6 will enroll adult subjects with cystic fibrosis on stable tezacaftor/ivacaftor background therapy. Approximately 104 subjects will be enrolled in Part 2.

DETAILED DESCRIPTION:
PART 1 The SAD treatment group is comprised of three cohorts where HV will be randomized to either PTI-801 or placebo. The MAD treatment group is comprised of three cohorts where subjects will be randomized to receive either PTI-801 or placebo once daily (QD) for a total of 7 days. HV will participate in a FE treatment group ,the FE treatment group is comprised of one cohort where subjects will be randomized to receive an initial single dose of PTI-801 either after an overnight fast of at least 10 hours (fasted group) or after an overnight fast of at least 10 hours followed by the consumption of a high fat high and high calorie meal (fed group). A set of HV will participate in a DDI treatment group. The DDI treatment group is comprised of one cohort where subjects will receive a 3-drug cocktail consisting of caffeine, bupropion, and midazolam on Day 1. On Day 4, subjects will be randomized to receive either PTI-801 or placebo QD for a total of 12 days. On Day 17, subjects will receive the 3-drug cocktail in combination with PTI-801 or placebo.

PART 2 Part 2 is comprised of a MAD treatment group with three cohorts, a co-administration group with two cohorts and a treatment group with one cohort.

Following the conclusion of the complementary HV MAD Cohort in Part 1, a set of adult subjects diagnosed with CF currently on a stable ivacaftor/lumacaftor background therapy for a minimum of three months will participate in the Part 2 complementary CF MAD cohort. Subjects will be randomized to receive either PTI-801 or placebo QD for a total of 14 days.

Following the conclusion of CF MAD Cohort 1 in Part 2, a set of adult subjects diagnosed with CF not currently receiving or have received background CFTR modulator therapy for a minimum of 30 days prior to Day 1 will participate in the Part 2 CF PTI-801 and PTI-808 co-administration cohort. Subjects will be randomized to receive either PTI-801 co-administered with PTI-808 or placebos QD for a total of 14 days.

Following the conclusion of the CF MAD Cohort 1 in Part 2, a set of adult subjects diagnosed with CF currently on a stable tezacaftor/ivacaftor background therapy for a minimum of one month will participate in the Part 2 complementary CF cohort. Subjects will be randomized to receive either PTI-801 or placebo QD for a total of 14 days.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Adults age 18 to 55 years old, inclusive, at the time of informed consent.
* Body mass index (BMI) ≥18 to <30 kg/m2.
* Subject must be a nonsmoker and a nontobacco user for a minimum of 30 days prior to screening and for the duration of the study.

Part 1 Exclusion Criteria:

* History or current evidence of any clinically significant cardiac, endocrinologic,hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic,dermatologic, psychiatric, renal, or other major disease, as determined by the investigator.
* Presence of prolonged QT/ Corrected QT Interval (QTc) interval with Fridericia's correction formula (QTcF) >450 msec at screening.
* Abnormal liver function as defined by aspartate aminotransferase (AST), alanine aminotransferase (ALT) or bilirubin > upper limit of the normal range.
* Abnormal renal function at screening defined as: Creatinine clearance <80 mL/min using the Cockcroft-Gault equation.
* Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to Study Day 1.
* History of cancer within the past 5 years (excluding nonmelanoma skin cancer).
* History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator.
* Positive urine screen for prohibited drugs (cocaine, cannabinoids, nicotine [urine cotinine is the detection mechanism for nicotine], opiates, barbiturates, amphetamines, and benzodiazepines) or positive alcohol test at screening.
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb).
* Has donated blood within 3 months of screening or plans to donate blood within 3 months of study completion.

Part 1 HV DDI Cohort Additional Exclusion Criteria:

* Concomitant use of known strong or moderate inhibitors or inducers of CYP1A2, CYP2B6, and CYP3A4 within 14 days or 5 half-lives (whichever is longer) prior to Day 1 and through the last PK sampling point on Day 20
* Use of grapefruit- or Seville orange-containing products within 48 hours prior to Day 1 and through the last PK sampling point on Day 20
* Use of alcohol- or caffeine-containing products within 48 hours prior to Day 1 and through the last PK sampling point on Day 20

Part 2 Inclusion Criteria:

* Confirmed diagnosis of CF with the F508del/F508del genotype on record, along with clinical findings consistent with CF such as chronic sinopulmonary disease or gastrointestinal/nutritional abnormalities
* Forced expiratory volume in 1 second (FEV1) 40-90% predicted, inclusive
* Non-smoker and non-tobacco user for a minimum of 30 days prior to screening

Part 2 Cohorts 1-3 Additional Inclusion Criterion:

* Stable on ivacaftor/lumacaftor dosing for both label indication and per label dosing for a minimum of 3 months at the time of dosing

Part 2 Cohort 6 Additional Inclusion Criterion:

* Stable on tezacaftor/ivacaftor dosing for both label indication and per label dosing for a minimum of 1 month at the time dosing

Part 2 Exclusion Criteria:

* Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Study Day 1
* History of cancer within the past 5 years (excluding cervical cancer in situ with curative therapy for at least one year prior to screening and non-melanoma skin cancer)
* History of organ transplantation
* Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (as determined by the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 14 days of Day 1
* Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®)) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to Day 1
* History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
* Pregnant or nursing women

Part 2 Cohort's 4 and 5 Additional Exclusion Criterion:

* Currently taking or has taken a CFTR modulator within 30 days prior to initial dose of study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Part 1 SAD and MAD HV: Safety and tolerability measured by number of subjects who experience adverse events and potential clinically significant changes in safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | baseline to up to 14 days
Part 1 SAD: Apparent terminal half-life (t1/2) of single oral dose | through 72-hours post dose
Part 1 SAD: Time to reach maximum plasma concentration (Tmax) of single oral dose | through 72-hours post dose
Part 1 SAD: Maximum plasma concentration (Cmax) of single oral dose | through 72-hours post dose
Part 1 SAD: Area under the concentration-time curve from time 0 to 24 hours post administration (AUC0-24) of a single oral dose | through 72-hours post dose
Part 1 SAD: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-last) of a single oral dose | through 72-hours post dose
Part 1 SAD: AUC from time 0 to infinity (AUC0-inf) | through 72-hours post dose
  using noncompartmental methods as appropriate of single dose
Part 1 MAD HV: Apparent terminal half-life (t1/2) of multiple oral doses | through 72-hours post last dose
Part 1 MAD HV: Time to reach maximum plasma concentration (Tmax) of multiple oral doses | through 72-hours post last dose
Part 1 MAD HV: Maximum plasma concentration (Cmax) of multiple oral doses | through 72-hours post last dose
Part 1 MAD HV: Area under the concentration-time curve from time 0 to 24 hours post administration (AUC0-24) of multiple oral doses | through 72-hours post dose
Part 1 MAD HV: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUClast) of multiple oral doses | through 72-hour post last dose
Part 1 MAD HV: AUC from time 0 to infinity (AUC0-inf) of multiple oral doses | through 72-hour post last dose
  using noncompartmental methods as appropriate of multiple oral doses
Part 1 MAD HV: Cumulative amount of PTI-801 excreted unchanged in urine (Ae) as appropriate of multiple oral doses | through 24-hour post last dose
Part 1 MAD HV: Cumulative amount of PTI-801 unchanged in renal clearance (CLR) as appropriate of multiple oral doses | through 24-hour post last dose
Part 1 FE: Time to reach maximum plasma concentration (Tmax) | through 72-hour post last dose
Part 1 FE :Maximum plasma concentration (Cmax) | through 72-hour post last dose
Part 1 FE: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUCt) | through 72-hour post last dose
Part 1 FE: AUC from time 0 to infinity (AUC0-inf) | through 72-hour post last dose
Part 1 DDI: Safety and tolerability measured by number of subjects who experience adverse events and potential clinically significant changes in safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | baseline through 7 days post last dose
Part 1 DDI: Maximum plasma concentration (Cmax) of caffeine, bupropion, and midazolam with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUClast) of caffeine, bupropion, and midazolam with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Area under the concentration-time curve from time 0 to infinity (AUCinf) of caffeine, bupropion, and midazolam with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 2 CF: Safety and tolerability measured by number of subjects who experience adverse events and potential clinically significant changes in safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | baseline through Day 21

SECONDARY OUTCOMES:
Part 1 FE: Safety and tolerability measured by number of subjects who experience adverse events and potential clinically significant changes in safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | baseline through 7 days post last dose
Part 1 DDI: Apparent terminal half-life (t1/2) of multiple oral doses of PTI-801 with and without caffeine, bupropion, and midazolam | through 72-hours post dose
Part 1 DDI: Time to reach maximum plasma concentration (Tmax) of the metabolites of caffeine, bupropion, and midazolam after single oral doses of caffeine, bupropion, midazolam, and with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Maximum plasma concentration (Cmax) of the metabolites of caffeine, bupropion, and midazolam after single oral doses of caffeine, bupropion, midazolam, and with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: AUClast of the metabolites of caffeine, bupropion, and midazolam after single oral doses of caffeine, bupropion, midazolam, and with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Area under the concentration-time curve from time 0 to 24 hours post administration (AUC0-24) of multiple oral doses of PTI-801 with and without caffeine, bupropion, and midazolam | through 72-hours post dose
Part 1 DDI: Metabolite over parent ratio of Cmax of single oral doses of the metabolites of caffeine, bupropion, and midazolam after single oral doses of caffeine, bupropion, midazolam, and with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Metabolite over parent ratio of AUClast of the metabolites of caffeine, bupropion, and midazolam after single oral doses of caffeine, bupropion, midazolam, and with and without multiple oral doses of PTI-801 | through 72-hours post dose
Part 1 DDI: Time to reach maximum plasma concentration (Tmax) of multiple oral doses of PTI-801 with and without caffeine, bupropion, and midazolam | through 72-hours post dose
Part 1 DDI: Maximum plasma concentration (Cmax) of multiple oral doses of PTI-801 with and without caffeine, bupropion, and midazolam | through 72-hours post dose
Part 1 DDI: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUClast) of multiple oral doses of PTI-801 with and without caffeine, bupropion, and midazolam | through 72-hours post dose
Part 2 CF: Time to reach maximum plasma concentration (Tmax) | Day 1 through Day 15
Part 2 CF: Maximum plasma concentration (Cmax) | Day 1 through Day 15
Part 2 CF: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUClast) | Day 1 through Day 15
Part 2 CF: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUClast) of multiple oral doses of PTI-808 with PTI-801 | Day 1 through Day 15
Part 2 CF: change in forced expiratory volume in one second (FEV1) over time | baseline through Day 21

OTHER OUTCOMES:
Part 1 SAD, MAD HV, and FE: The effect of PTI-801 on the QT interval as measured by holter monitoring | baseline through 7 days post last dose
Part 1: change in nasal epithelial mRNA and protein expression over time | baseline through 7 days post last dose
Part 2 CF: change in sweat chloride over time | baseline through Day 21
Part 2 CF: change in nasal epithelial mRNA and protein expression over time | baseline through Day 21
Part 2 CF: change in weight and BMI over time | baseline through Day 21
Part 2 CF: change in blood glucose over time | baseline through Day 21

CONTACTS AND LOCATIONS:
Locations (38):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami Health System, Miami, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Children's Mercy Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Children's Lung Specialists, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Mount Sinai Beth Israel, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Health System, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Santiago Reyes, M.D. P.C., Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - ICON Early Phase Services, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- University of Copenhagen Rigshospitalet, Copenhagen, Denmark
- Charite - Campus Virchow-Klinikum, Berlin, Germany
- Stockholm CF Center, Stockholm, Sweden